CLINICAL TRIAL: NCT01917929
Title: A Prospective, Post-market, Multi-center Evaluation of the Clinical Outcomes of the Secur-Fit Advanced Hip Stem
Brief Title: Secur-Fit Advanced Outcomes Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As longitudinal patient follow up continues to lag, Stryker has determined that the study is no longer able to meet the regulatory requirements it was intended to support. Termination is not related to any safety concerns with the product.
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 75
Record Dates: First submitted 2013-06-24; First posted 2013-08-07 (Estimated); Results first posted 2024-11-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: [E04.555.110.110.110]

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Secur-Fit Advanced (Other): Secur-Fit Advanced Hip Stem
  Interventions: Device: Secur-Fit Advanced Hip Stem

INTERVENTIONS:
Device: Secur-Fit Advanced Hip Stem — Straight femoral stem intended for cementless, press-fit application.

SUMMARY:
The goal of this study is to evaluate the Secur-Fit Advanced Hip Stem in primary total hip replacement surgery.

DETAILED DESCRIPTION:
This study is a prospective, open-label, post-market, non-randomized, multi-center clinical evaluation of the Secur-Fit Advanced Hip Stem for primary total hip arthroplasty with a cementless application in a consecutive series of patients who meet the eligibility criteria.

The primary objective of this study is to evaluate the success rate of cementless primary total hip replacement with the Secur-Fit Advanced Hip Stem. Success will be defined as absence of femoral stem revision for aseptic loosening or device-related femoral fracture at 5 years postoperative. It is expected that the success rate of the Secur-Fit Advanced Hip Stem group will be non-inferior to the selected reference rate of 99% at 5 years postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed an Institutional Review Board (IRB)/Ethics Committee (EC) approved, study specific Informed Patient Consent Form.
* Patient is a male or non-pregnant female, skeletally mature and age 21-75 years at time of study device implantation.
* Patient has a diagnosis of Non-Inflammatory Degenerative Joint Disease.
* Patient is a candidate for primary total hip arthroplasty.
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* Patient has previously undergone open surgical intervention on the operative hip.
* Patient has a prior femoral fracture, with or without deformity, on the operative side.
* Patient has an existing total hip replacement on the contralateral side.
* Patient requires simultaneous bilateral total hip replacement.
* Patient has a Body Mass Index (BMI) > 45.
* Patient has an active or suspected latent infection in or about the affected hip joint at time of study device implantation.
* Patient has a neuromuscular or neurosensory deficiency that would create an unacceptable risk of instability, prosthesis fixation failure or complications in postoperative care, or which limits the ability to evaluate the safety and efficacy of the device.
* Patient has bone stock that is inadequate for support or fixation of the prosthesis, or is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's disease) leading to progressive bone deterioration.
* Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
* Patient has a known sensitivity to device materials.
* Patient is a prisoner.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2013-08-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Petrow, MD, Principal Investigator — Tucson Orthopaedic Institute; Geoffrey Westrich, MD, Principal Investigator — Hospital for Special Surgery, New York; Samuel Wellman, MD, Principal Investigator — Duke University; Paul Perona, MD, Principal Investigator — Family Orthopaedic Center; Michael Dayton, MD, Principal Investigator — University of Colorado, Denver; Thomas Bowen, MD, Principal Investigator — Geisinger Orthopaedic Institute; Frank Conguista, MD, Principal Investigator — Ortho NY; Michael Ast, MD, Principal Investigator — Mercer Bucks Orthopaedics
Locations (8):
- United States (8):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - University of Colorado Denver, Aurora, Colorado
  - Family Orthopedic Center, Spring Valley, Illinois
  - Mercer Bucks Orthopaedics, Lawrenceville, New Jersey
  - OrthoNY - Everett Road Health Park, Albany, New York
  - Hospital for Special Surgery, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Geisinger Orthopaedic Institute, Danville, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 326 hips/participants enrolled in this study (no bilateral cases).
Pre-assignment Details: Of the 326 hips/participants enrolled and consented, there were 12 cases that were censored due to not having the study device implanted, surgery cancelled or due to an inclusion or exclusion violation. Therefore, 314 hips/participants (there were no bilateral cases) are followed who did receive the study device and met protocol criteria. Those applicable data are reflected in this record.
Period: Overall Study
Arm/Group | Secur-Fit Advanced
Started | 326
Completed | 38
Not Completed | 288
Not completed — Death | 8
Not completed — Lost to Follow-up | 19
Not completed — Withdrawal by Subject | 33
Not completed — Adverse Event | 6
Not completed — Investigative Site Terminated | 35
Not completed — Censored because study device not implanted | 6
Not completed — Censored because surgery not performed | 3
Not completed — Censored because of inclusion exclusion violation | 3
Not completed — Sponsor terminated study | 175

BASELINE CHARACTERISTICS:
Arm/Group | Secur-Fit Advanced
Number analyzed (Participants) | 314
Age, Continuous [Mean (Full Range); unit: years] | 61.81 [32 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 163
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 286
  More than one race | 3
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Revision for Aseptic Loosening or Device-related Femoral Fracture
Description: The primary objective is to determine the success rate at 5 years postoperative with the Secur-Fit Advanced Hip Stem in the cementless application. Success is defined as absence of femoral stem revision and/or removal for aseptic loosening or device-related femoral fracture at 5 years postoperative.
Time Frame: 5 years
Population: Participants/hips with available data up to 5 years or at the time of early study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Secur-Fit Advanced
Number analyzed (Participants) | 314
Participants | 0

2. Secondary Outcome: All-cause Revision and Removal Rate
Description: To evaluate all-cause revision and removal rates with the Secur-Fit Advanced Hip Stem and compare with those reported for other primary hip stems in the literature.
Time Frame: 10 years
Population: Participants/hips with available data up to 10 years or at the time of early study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Secur-Fit Advanced
Number analyzed (Participants) | 314
Participants | 6

3. Secondary Outcome: Rate of Device-related Femoral Fracture
Description: To evaluate rate of device-related femoral fracture among patients implanted with the Secur-Fit Advanced Hip Stem within 30 days postoperative, and compare with rates reported for other primary hip stems in the literature.
Time Frame: 30 days
Population: Participants/hips with available data from surgery to 30 days postoperative.
Measure: Count of Participants; unit: Participants
Arm/Group | Secur-Fit Advanced
Number analyzed (Participants) | 314
Participants | 1

4. Secondary Outcome: Final Seating of Femoral Stem
Description: To demonstrate the close relationship between the seating height of the Secur-Fit Advanced Hip Stem and its associated femoral broach by intraoperatively measuring the component exposure or countersink upon final seating.
Time Frame: Intraoperative
Population: Participants/hips with available data intraoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Secur-Fit Advanced
Number analyzed (Participants) | 314
Participants
  Flush seating on femoral stem | 223
  Proud seating of femoral stem | 82
  Countersunk seating of femoral stem | 9

ADVERSE EVENTS:
Time Frame: The study period during which the AEs must be reported is defined as the period from the initiation of any study procedures to the end of the study treatment follow-up at 10-years or study closure. The start of study procedures is considered to be the date of consent. Any AEs that met the protocol defined reportable events were required to be reported from the time of consent until study completion.
Description: Serious systemic adverse events that occurred within the perioperative period (intraoperative to hospital discharge) were required to be reported.
  All operative site events, regardless of seriousness or time of occurrence were required to be reported.
Groups:
- Operative Site Events: All adverse events whether serious or not that occurred within the study population of 314 participants/hips (there were no bilateral cases).
- Non Operative Site Events (Systemic): All serious systemic adverse events that occurred in the study population in the perioperative period (intraoperative to hospital discharge) in 314 participants/hips.
Arm/Group | Operative Site Events | Non Operative Site Events (Systemic)
All-Cause Mortality (participants affected / at risk) | 0/314 | 8/314
Serious Adverse Events (participants affected / at risk) | 14/314 | 4/314
Other Adverse Events (participants affected / at risk) | 27/314 | 0/314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative Site Events (N=314) | Non Operative Site Events (Systemic) (N=314)
Systemic Other (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Acute blood loss anemia
Urogenital (Renal and urinary disorders) | 0 (0) | 1 (1)
Systemic Other (Surgical and medical procedures) | 0 (0) | 1 (1) — Acute blood loss anemia
Deep Joint Infection (Infections and infestations) | 1 (1) | 0 (0)
Superficial Wound Infection (Infections and infestations) | 2 (2) | 0 (0)
Femoral Crack (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femoral Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Femoral Component Subsidence (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Femoral Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Operative Site Other (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Metallosis from stem/cup impingement
Operative Site Other (Surgical and medical procedures) | 1 (1) | 0 (0) — Elevated chromium and cobalt levels
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative Site Events (N=314) | Non Operative Site Events (Systemic) (N=314)
Bursitis (Musculoskeletal and connective tissue disorders) | 27 (29) | 0 (0)

LIMITATIONS AND CAVEATS:
Given the challenges initiated by the COVID-19 pandemic and the difficulties in recalling study subjects for long-term postoperative visits, follow-up compliance saw a decline. As a result, the number of subjects available for analysis at the 10-year endpoint would be insufficient. Consequently, a business decision was made to close the study early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each study investigator has independent publication privileges for their own center's results after multi-center publications are submitted. Sponsor requires review of publications. Sponsor shall not edit or influence the publications except to ensure that confidential information is not disclosed, no off-label device use is promoted, and that data is accurately represented. Any publications must be submitted to Stryker for review at least 60 days prior to submission of publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT01917929/Prot_SAP_000.pdf